CLINICAL TRIAL: NCT03100838
Title: A Single-Dose, Open-label, Randomized, Crossover, Drug-Drug Interaction Study of Nifedipine Extended-release Tablets With or Without Multiple-dose Administration of Proton-Pump Inhibitor Omeprazole/Sodium Bicarbonate in Healthy Volunteers
Brief Title: Drug Interaction With Proton Pump Inhibitors for Nifedipine ER Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: BioPharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RIHSC 16-070D
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers
Keywords: Proton Pump Inhibitor; Bioequivalence; Drug-Drug Interaction; Modified Release; Nifedipine
MeSH Terms: interventions — Nifedipine; omeprazole, sodium bicarbonate drug combination

STUDY DESIGN:
Intervention Model Description: A single-dose, randomized, open-label, drug-drug interaction (DDI), 4-way crossover, four-treatment, four-sequence, bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nifedipine (Generic) (Experimental): 1 x 60 mg Nifedipine extended-release tablet
  Interventions: Drug: Nifedipine 60 MG Extended Release Oral Tablet; Device: SmartPill (TM)
- Nifedipine (Brand) (Active Comparator): 1 x 60 mg PROCARDIA XL (nifedipine) extended-release tablet
  Interventions: Drug: Nifedipine 60 MG Extended Release Oral Tablet; Device: SmartPill (TM)
- Nifedipine (Generic) + PPI (Active Comparator): 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 7 days + 1 x 60 mg Nifedipine extended-release tablet on day 7
  Interventions: Drug: Nifedipine 60 MG Extended Release Oral Tablet; Drug: omeprazole/sodium bicarbonate; Device: SmartPill (TM)
- Nifedipine (brand) + PPI (Active Comparator): 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 7 days + 1 x 60 mg PROCARDIA XL (nifedipine) extended-release tablet on day 7
  Interventions: Drug: Nifedipine 60 MG Extended Release Oral Tablet; Drug: omeprazole/sodium bicarbonate; Device: SmartPill (TM)

INTERVENTIONS:
Drug: Nifedipine 60 MG Extended Release Oral Tablet — Reference Drug (Brand)
  Other Names: Procardia XL
  Arms: Nifedipine (Brand); Nifedipine (brand) + PPI
Drug: Nifedipine 60 MG Extended Release Oral Tablet — Test Drug (Generic)
  Arms: Nifedipine (Generic); Nifedipine (Generic) + PPI
Drug: omeprazole/sodium bicarbonate — Proton Pump Inhibitor/Antacid for drug-drug interaction
  Arms: Nifedipine (Generic) + PPI; Nifedipine (brand) + PPI
Device: SmartPill (TM) — Gastric pH measurement using SmartPill (TM) Technology

SUMMARY:
The purpose of this study is to measure the amount of study drug present in blood after being administered a generic version of nifedipine extended-release tablets, 60 mg (Valeant Pharmaceuticals, LLC) and brand-name version PROCARDIA XL extended-release tablets, 60 mg (Pfizer Inc.) individually and in presence of stomach acid reducing drug (antacid), omeprazole/sodium bicarbonate capsules, 40 mg/1100 mg (generic) on separate occasions, on an empty stomach. This study also involves administrations of an FDA-cleared capsule, SmartPill™, which will measure stomach acid, prior to each study arm.

DETAILED DESCRIPTION:
A question that arises with generic oral extended-release (ER) products is related to pH-dependent dissolution kinetics in comparison with that of their reference listed drug (RLD). For example, poorly water-soluble drugs with the presence of pKa in the gastrointestinal (GI) pH range have pH-dependent solubility and dissolution behaviors during in vivo drug release. In this case, the generic product which utilizes a different release mechanism could amplify or reduce such a pH dependence (e.g. osmotic pump RLD vs. matrix generic counterparts). This may render these generic ER products more or less dependent on gastric pH modification, commonly occurred in patients taking concomitant over-the-counter (OTC) proton pump inhibitors (PPIs) for the treatment of gastric acid-related disorders. It has been noted that PPIs (e.g. lansoprazole, omeprazole, esomeprazole) and PPIs with antacids (e.g. omeprazole/sodium bicarbonate) can drastically elevate the gastric pH, thus potentially changing the equilibrium solubility of co-administered drug substances or altering their release profiles.

For instance, nifedipine is a calcium channel blocker, indicated for the long-term treatment of hypertension and angina. The drug substance is a weak acid (pKa 3.9) and practically insoluble in water. Currently, there is one RLD of oral ER nifedipine tablets based on an osmotic pump design (Procardia XL) and a generic counterpart of ER nifedipine tablets employing a matrix formulation design which is different from this RLD product. Due to complicated release mechanisms, quality attribute profiles, and in vivo pharmacokinetics (PK) behaviors of ER products, FDA is assessing the need of a drug-drug interaction study between PPIs/antacids (e.g. omeprazole/sodium bicarbonate) and generic nifedipine ER products based on a formulation design which is different from that of its RLD.

To this end, the objective of this proposal is to investigate the dependence of in vivo PK on the formulation design of generic oral extended-release products in comparison with that of their RLD when co-administered with PPIs/antacids. The outcome of this study will help the Agency advance further understanding about product PK performance in potential patient population with abnormal gastric pH and improve review standards for equivalence of this category of oral ER products if necessary. The study results will help the Agency gain a better understanding of drug-drug interaction between oral modified-release products and PPIs/antacids and establish regulatory standards of bioequivalence approaches for this category of generic oral ER products.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, males and non-pregnant female volunteers, 18 to 55 years of age, inclusive.
2. Smoking status: Only non-tobacco/nicotine users (for at least 6 months prior to the clinical study) will be eligible to participate in this study.
3. BMI that is within 18.5-35.0 kg/m², inclusive.
4. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
5. Ability to comprehend and be informed of the nature of the study, as assessed by BPSI staff. Capable of giving written informed consent prior to receiving any study procedure. Must be able to communicate effectively with clinic staff.
6. Ability to fast for at least 14 hours.
7. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
8. Female subjects must fulfill at least one of the following:

   * Be surgically sterile for a minimum of 6 months;
   * Post-menopausal for a minimum of 1 year;
   * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study until 30 days after the study has ended (last study procedure).

Medically acceptable methods of contraception include non-hormonal contraceptives, intrauterine device, or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicide). Complete abstinence alone can be used as a method of contraception.

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal (e.g., gastrointestinal obstruction, gastrointestinal ulcers), cardiovascular (e.g., severe obstructive coronary artery disease, myocardial infarction, angina, heart failure), cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting, swallowing disorder), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first dosing, as determined by the PI/Sub-Investigator.
3. QTc interval > 430 milliseconds for males and > 450 milliseconds for females, unless deemed otherwise by the PI/Sub-Investigator.
4. Abnormal clinical laboratory values, unless values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".
5. Hemoglobin values less than 11.5 g/dl.
6. Abnormal vital signs (blood pressure [BP], heart rate [HR], respiratory rate [RR] and temperature) measurements, unless deemed otherwise by the PI/Sub-Investigator.
7. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
8. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
9. Individuals who have implanted or portable electro-mechanical medical device such as a cardiac pacemaker, defibrillator or infusion pump.
10. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol test and cotinine. Positive pregnancy test for female subjects.
11. Known history or presence of:

    * Alcohol abuse or dependence within one year prior to first study period;
    * Drug abuse or dependence;
    * Hypersensitivity or idiosyncratic reaction to nifedipine, omeprazole/sodium bicarbonate, its excipients, and/or related substances;
    * Hypotension;
    * Bartter's syndrome;
    * Gastric bezoar;
    * Crohn's disease or diverticulitis;
    * severe dysphagia to food or pills;
    * Food allergies and/or presence of any dietary restrictions;
    * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
12. History of intolerance to and/or difficulty with blood sampling through venipuncture.
13. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets, vegan, etc.
14. Individuals who have donated, in the days prior to first study period:

    * 50-499 mL of blood in the previous 30 days;
    * 500 mL or more in the previous 56 days.
15. Donation of plasma by plasmapheresis within 7 days prior to first study period.
16. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study period.
17. Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g. cimetidine, fluoxetine, quinidine, fluconazole, ketoconazole, voriconazole, itraconazole, clarithromycin, erythromycin, nefazodone, atazanavir, saquinavir, indinavir, and nelfinavir) and strong inducers of CYP enzymes (e.g. barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort and rifampin) in the previous 30 days before first study period.
18. Use of drugs such as, proton pump inhibitors, clopidogrel, tacrolimus, digoxin, cyclosporine, disulfiram, benzodiazepines, diazepam, warfarin, methotrexate, iron salts, erlotinib, and mycophenolate mofetil (MMF) in the previous 30 days before first study period, or individuals with vitamin B-12 deficiency (as long-term dosing (more than 3 years) of omeprazole/sodium bicarbonateZegerid may lead to vitamin B-12 deficiency)
19. Individuals having undergone gastrointestinal (GI) surgery within 3 months prior to first study period, unless deemed otherwise by PI/Sub-Investigator.
20. Use of any prescription medication within 14 days prior to first study period (except for contraceptives).
21. Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements and/or teas) within 14 days prior to first study period (except for spermicidal/barrier contraceptive products).
22. Consumption of food or beverages containing grapefruit and grapefruit juice and/or pomelo within 10 days prior to first study period.
23. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing.
24. Use of diuretics (drugs or food, see Appendix D) within 24 hours before dosing of SmartPillTM.
25. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
26. Difficulty with swallowing whole tablets or large capsules.
27. Have had a tattoo or body piercing within 30 days prior to first study period and during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2018-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Doisy, Principal Investigator — BioPharma Inc.
Locations (1):
- BioPharma Services Inc., Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have the plans to share the de-identified IPD at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 subjects were dosed.
Groups:
- Sequence 1 (ABCD); Sequence 2 (BCDA); Sequence 4 (DABC): A Generic 1 x 60 mg Nifedipine extended-release tablet
  B Brand (Procardia XL)
  1 x 60 mg Nifedipine extended-release tablet
  C Generic+PPI (antacids) 1 x 60 mg Nifedipine extended-release tablet 7 x 40 mg omeprazole/1100 mg sodium bicarbonate capsules
  D Brand (Procardia XL) +PPI (antacids)
  1 x 60 mg Nifedipine extended-release tablet 7 x 40 mg omeprazole/1100 mg sodium bicarbonate capsules
  A washout period of at least 14 days occurs between each intervention.
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
- Sequence 3 (CDAB): A Generic 1 x 60 mg Nifedipine extended-release tablet
  B Brand (Procardia)
  1 x 60 mg Nifedipine extended-release tablet
  C Generic+PPI (antacids) 1 x 60 mg Nifedipine extended-release tablet 7 x 40 mg omeprazole/1100 mg sodium bicarbonate capsules
  D Brand (Procardia) +PPI (antacids)
  1 x 60 mg Nifedipine extended-release tablet 7 x 40 mg omeprazole/1100 mg sodium bicarbonate capsules
  A washout period of at least 14 days occurs between each intervention.
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
Period: Overall Study
Arm/Group | Sequence 1 (ABCD) | Sequence 2 (BCDA) | Sequence 3 (CDAB) | Sequence 4 (DABC)
Started | 16 | 16 | 16 | 16
Completed | 14 | 14 | 14 | 15
Not Completed | 2 | 2 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 1 | 1
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study. There are 64 subjects enrolled, but only 59 completed at least two treatments.
Groups:
- All Participants: Participants were randomized to one of the four sequences and were to receive all interventions.
Arm/Group | All Participants
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 32
  White | 21
  More than one race | 0
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Measurement of plasma nifedipine prior to dosing and at times 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 20, 24, 36 and 48 hr after nifedipine administration.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Nifedipine (Generic): 1 x 60 mg Nifedipine extended-release tablet
  NIFEdipine 60 MG: Test Drug
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
- Nifedipine (Brand): 1 x 60 mg PROCARDIA XL (nifedipine) extended-release tablet
  NIFEdipine 60 MG: Reference Drug
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
- Nifedipine (Generic) + PPI: 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 7 days + 1 x 60 mg Nifedipine extended-release tablet on day 7
  NIFEdipine 60 MG: Test Drug
  omeprazole/sodium bicarbonate: Proton Pump Inhibitor/Antacid for drug-drug interaction
- Nifedipine (Brand) + PPI: 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 7 days + 1 x 60 mg PROCARDIA XL (nifedipine) extended-release tablet on day 7
  NIFEdipine 60 MG: Reference Drug
  omeprazole/sodium bicarbonate: Proton Pump Inhibitor/Antacid for drug-drug interaction
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
Number analyzed (Participants) | 59 | 59 | 57 | 55
ng/mL | 94.37 (42.42) | 43.84 (44.07) | 106.35 (43.67) | 51.65 (32.47)

2. Primary Outcome: Time at Maximum Plasma Concentration (Tmax)
Description: as for outcome 1
Time Frame: 48 hours
Measure: Mean (Full Range); unit: hr
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
Number analyzed (Participants) | 59 | 59 | 59 | 59
hr | 4 [2 to 16] | 16 [3 to 36] | 6 [3 to 24] | 16 [5 to 36.02]

3. Primary Outcome: Area Under the Concentration (AUC 0-t)
Description: Time curve from time zero to last measurable concentration. Measurement of plasma nifedipine prior to dosing and at times 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 20, 24, 36 and 48 hr after nifedipine administration.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
Number analyzed (Participants) | 59 | 59 | 59 | 59
ng.h/mL | 1166.21 (45.64) | 1061.49 (47.52) | 1514.83 (29.95) | 1239.26 (40.68)

4. Primary Outcome: Half-life
Description: The apparent terminal exponential half-life. Measurement of plasma nifedipine prior to dosing and at times 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 20, 24, 36 and 48 hr after nifedipine administration.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
Number analyzed (Participants) | 59 | 59 | 59 | 59
hr | 8.59 (33.15) | 11.29 (82.39) | 8.10 (32.64) | 12.71 (119.78)

5. Secondary Outcome: Adverse Events
Description: Reported from the start of the first session to the follow-up visit.
Time Frame: 66 days
Measure: Number; unit: Events
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
Number analyzed (Participants) | 59 | 59 | 59 | 59
Events | 37 | 19 | 51 | 38

ADVERSE EVENTS:
Time Frame: Approximately 2 months
Groups:
- Nifedipine (Generic) + PPI: 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 8 days + 60 mg Nifedipine extended-release tablet on day 7
  NIFEdipine 60 MG: Test Drug
  omeprazole/sodium bicarbonate: Proton Pump Inhibitor/Antacid for drug-drug interaction
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
- Nifedipine (Brand) + PPI: 1 x 40 mg/1100 mg omeprazole/sodium bicarbonate capsule daily over a period of 8 days + 60 mg PROCARDIA XL (nifedipine) extended-release tablet on day 7
  NIFEdipine 60 MG: Reference Drug
  omeprazole/sodium bicarbonate: Proton Pump Inhibitor/Antacid for drug-drug interaction
  SmartPill (TM): Gastric pH measurement using SmartPill (TM) Technology
Arm/Group | Nifedipine (Generic) | Nifedipine (Brand) | Nifedipine (Generic) + PPI | Nifedipine (Brand) + PPI
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 23/59 | 15/59 | 38/59 | 28/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nifedipine (Generic) (N=59) | Nifedipine (Brand) (N=59) | Nifedipine (Generic) + PPI (N=59) | Nifedipine (Brand) + PPI (N=59)
Headache (Nervous system disorders) | 20 | 14 | 25 | 22
Constipation (Gastrointestinal disorders) | 1 | 1 | 5 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03100838/Prot_SAP_000.pdf